CLINICAL TRIAL: NCT04204603
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2a Study Investigating the Efficacy, Safety, Pharmacokinetic and Biomarker Profiles of CKD-506 Administered to Adult Subjects With Moderate-to- Severe Rheumatoid Arthritis and Inadequate Response to Methotrexate
Brief Title: A Study Evaluating the Efficacy and Safety of CKD-506 in Adult Subjects With Moderate-to-Severe Rheumatoid Arthritis and Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 182RA18009
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CKD-506

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CKD-506 Dose A (Experimental)
  Interventions: Drug: CKD-506
- CKD-506 Dose B (Experimental)
  Interventions: Drug: CKD-506
- CKD-506 Dose C (Experimental)
  Interventions: Drug: CKD-506

INTERVENTIONS:
Drug: CKD-506 — Tablets for oral administration
  Arms: CKD-506 Dose A; CKD-506 Dose B; CKD-506 Dose C
Drug: Placebo — Tablets for oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effects of CKD-506 on signs and symptoms of RA in subjects with moderate-to-severe RA who are inadequate responders to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for at least 6 months prior to Screening, currently meet the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria for RA, and are ACR functional class I-III.
* Have active RA
* Ongoing treatment with a stable dose of MTX as described below:

  1. Use of oral or injectable MTX on a continuous basis for at least 12 weeks prior to Baseline and on a stable dose and route of administration between 15 mg and 25 mg/weekly for at least 8 weeks prior to Baseline and planned during the study.
  2. Subjects should be on an adequate and stable dose of folic acid for at least 4 weeks prior to first administration of study treatment and planned during the study.
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for at least 12 weeks after the last dose of study treatment.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and urine pregnancy test at Baseline
* Sexually active men, if not surgically sterile, must agree to use a medically acceptable form of contraception during the study and continue its use for at least 12 weeks after the last dose of study treatment.

Exclusion Criteria:

* Treatments for RA as follows: JAK inhibitors at any time; use of any currently licensed biologics with DMARD properties at any time.
* Use of oral steroids at a dose >10 mg/day of prednisone or prednisone equivalent or at a dose that has not been stable for at least 4 weeks prior to Screening.
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) which have not been at a stable dose or route of administration for at least 2 weeks prior to Baseline and planned during the study.
* History of tuberculosis (TB) infection.
* Positive serology for human immunodeficiency virus 1 or 2, hepatitis B virus or hepatitis C virus.
* Currently active infection or history of infection within the last 2 weeks of Screening or Baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in DAS28(CRP) at week 12 | Baseline and week 12

SECONDARY OUTCOMES:
Response to treatment based on the American College of Rheumatology 20% response criteria (ACR20) at Weeks 2, 4, 8, and 12 | At weeks 2, 4, 8 and 12
Change from Baseline in DAS28(CRP) at Weeks 2, 4, and 8 | Baseline and up to week 8
Response to treatment based on the ACR50 criteria at Weeks 2, 4, 8, and 12 | At weeks 2, 4, 8 and 12
Response to treatment based on the ACR70 criteria at Weeks 2, 4, 8, and 12 | At weeks 2, 4, 8 and 12
Change from Baseline in ACRn at Weeks 2, 4, 8, and 12 | Baseline and up to week 12
Change from Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) at Weeks 4 and 12 | Baseline and weeks 4, 12
Change from Baseline in the duration of morning stiffness (in minutes and in severity as measured with a visual analog scale [VAS]) at Weeks 2, 4, 8, and 12 | Baseline and up to week 12
  Morning stiffness severity was determined by the Patient's Assessment of Severity and Duration of Morning Stiffness questionnaire. Participants rated the severity of morning stiffness on awakening over the past 7 days on a scale from 0 (No morning stiffness) to 10 (Worst possible morning stiffness).
Change from Baseline in the Short Form-36 item Health Survey (SF-36) at Weeks 4 and 12 | Baseline and weeks 4, 12
  The Short Form-36 item Health Survey (SF-36) consists of eight scaled scores; physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. which are the weighted sums of the questions in their section. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Change from Baseline in the Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 8, and 12 | Baseline and up to week 12
Change from Baseline in the Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 8, and 12 | Baseline and up to week 12
Response to treatment based on the achievement of Low Disease Activity (LDA) status based on each of the following definitions at Weeks 2, 4, 8,and 12: DAS28(CRP) ≤ 3.2, SDAI ≤ 11.0, CDAI ≤ 10.0 at Weeks 2, 4, 8, and 12 | At weeks 2, 4, 8 and 12
Response to treatment based on the achievement of remission based on each of the following definitions at Weeks 2, 4, 8, and 12: DAS28(CRP) < 2.6, Boolean parameters, SDAI ≤ 3.3, CDAI ≤ 2.8 at Weeks 2, 4, 8, and 12 | At weeks 2, 4, 8 and 12
Improvement of physical ability defined as change from Baseline in HAQ-DI ≥ 0.22 at Weeks 2, 4, 8, and 12 | Baseline and up to week 12

CONTACTS AND LOCATIONS:
Locations (38):
- Czechia (8):
  - 182RA18009 Stie# CZ06, Broumov
  - 182RA18009 Stie# CZ03, Olomouc
  - 182RA18009 Stie# CZ02, Prague
  - 182RA18009 Stie# CZ05, Prague
  - 182RA18009 Stie# CZ07, Prague
  - 182RA18009 Stie# CZ08, Prague
  - 182RA18009 Stie# CZ09, Prague
  - 182RA18009 Stie# CZ01, Uherské Hradiště
- Georgia (4):
  - 182RA18009 Stie# UA03, Lviv
  - 182RA18009 Stie# GE01, Tbilisi
  - 182RA18009 Stie# GE02, Tbilisi
  - 182RA18009 Stie# GE03, Tbilisi
- Poland (10):
  - 182RA18009 Stie# PL04, Bydgoszcz
  - 182RA18009 Site# PL01, Elblag
  - 182RA18009 Stie# PL03, Grodzisk Mazowiecki
  - 182RA18009 Stie# PL02, Katowice
  - 182RA18009 Stie# PL07, Lodz
  - 182RA18009 Stie# PL06, Poznan
  - 182RA18009 Stie# PL08, Poznan
  - 182RA18009 Stie# PL05, Skierniewice
  - 182RA18009 Stie# PL10, Torun
  - 182RA18009 Stie# PL09, Warsaw
- Russia (8):
  - 182RA18009 Stie# RF05, Moscow
  - 182RA18009 Stie# RF10, Moscow
  - 182RA18009 Stie# RF09, Perm
  - 182RA18009 Stie# RF03, Saint Petersburg
  - 182RA18009 Stie# RF08, Saint Petersburg
  - 182RA18009 Stie# RF02, Tolyatti
  - 182RA18009 Stie# RF07, Tver'
  - 182RA18009 Stie# RF06, Vladimir
- Ukraine (8):
  - 182RA18009 Stie# UA10, Ivano-Frankivsk
  - 182RA18009 Stie# UA09, Kharkiv
  - 182RA18009 Stie# UA01, Kyiv
  - 182RA18009 Stie# UA04, Kyiv
  - 182RA18009 Stie# UA07, Kyiv
  - 182RA18009 Stie# UA11, Kyiv
  - 182RA18009 Stie# UA05, Vinnytsia
  - 182RA18009 Stie# UA06, Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided